CLINICAL TRIAL: NCT01039025
Title: Phase II Study of High-Dose Topotecan, Cyclophosphamide and Melphalan for the Treatment of Multiple Myeloma
Brief Title: TMC (Topotecan, Cyclophosphamide and Melphalan) for Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: SmithKline Beecham (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM01-331
Record Dates: First submitted 2009-12-23; First posted 2009-12-24 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Myeloma
Keywords: Myeloma; Topotecan; Hycamtin; Melphalan; Alkeran; Cyclophosphamide; Cytoxan; Neosar; Stem Cell Harvest; Peripheral Blood Stem Cells
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — Topotecan; Cyclophosphamide; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TMC (Experimental): Topotecan, Melphalan, and Cyclophosphamide
  Interventions: Drug: Topotecan; Drug: Cyclophosphamide; Drug: Melphalan; Other: Peripheral Blood Stem Cells

INTERVENTIONS:
Drug: Topotecan — After stem cells are collected, Topotecan 3.5 mg/m^2 intravenously given over 30 minutes on Days 1 - 5.
  Other Names: Hycamtin
Drug: Cyclophosphamide — After stem cells are collected, Cyclophosphamide 1 g/m^2/day intravenously given over 2 hours on Days 1 - 3.
  Other Names: Cytoxan; Neosar
Drug: Melphalan — After stem cells are collected, Melphalan 70 mg/m^2/day intravenously given on Days 4 and 5.
  Other Names: Alkeran
Other: Peripheral Blood Stem Cells — On Day 7, some or all of the stem cells will be reinfused.

SUMMARY:
To determine the efficacy of high-dose topotecan, cyclophosphamide and melphalan in patients with Multiple Myeloma.

DETAILED DESCRIPTION:
Patients in this study will have a catheter (a tube) placed in the vein below the collarbone. Most of the drugs used in the study will be given through the catheter. Blood stem cells will be collected through this tube also.

Before treatment starts, patients will have a complete physical exam, including blood and urine tests. A dentist will perform a dental exam either at M.D. Anderson or elsewhere. A chest x-ray and bone x-rays will be done. An EKG and a heart scan will be done to test heart function. A breathing test will be done. Patients will also be screened for HIV and Hepatitis.

Blood stem cells will be collected from patients when white blood cell counts are normal. This will be after earlier chemotherapy or after a bone marrow growth factor (G-CSF) has been given. Collecting stem cells takes about 3 hours. It takes from 1 to 6 sessions to get the needed amount of cells. The process is called apheresis. A machine is attached to the catheter, and blood is drawn. The machine removes the stem cells from the blood and the blood is then returned to the body through the catheter. G-CSF is injected under the skin twice a day during the time the stem cells are collected. The stem cells are stored frozen and will be used later to help patients recover from the high-dose chemotherapy.

After stem cells are collected, patients will receive high-dose chemotherapy. Cyclophosphamide is given over 2 hours on Days 1 - 3. Melphalan is given on Days 4 and 5. Topotecan is given over 30 minutes on Days 1 - 5, right after cyclophosphamide or melphalan. On Day 6, no drugs are given. On Day 7, some or all of the stem cells will be reinfused. G-CSF will be given once a day until blood counts return to normal.

Patients must stay in the hospital for the high-dose drug treatment. The length of stay will be about 3 weeks. Blood tests will be done daily while in hospital, then once a week for the first month. A bone marrow sample will be taken on Day 30. Blood samples will be taken 4 times in the first year and once a year after that. Thyroid gland tests and a bone marrow test will be done once a year.

This is an investigational study. Cyclophosphamide, melphalan, and topotecan are approved by the FDA. Their use together in this study is experimental. All participants will be enrolled at UTMDACC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with intermediate or high tumor mass multiple myeloma with responsive or primary refractory disease; and patients with responsive or refractory relapse.
2. Physiological age </= 70.
3. Zubrod performance status < 3.
4. Life expectancy greater than 12 weeks.
5. Left ventricular ejection fraction >/= 50%.
6. No uncontrolled arrythmias or symptomatic cardiac disease.
7. FEV1, FVC and DLCO >/= 50%.
8. No symptomatic pulmonary disease.
9. Serum creatinine < 1.5 mg/dL.
10. Serum bilirubin < 2x upper limit of normal.
11. No evidence of chronic or active hepatitis or cirrhosis.
12. Patient is not pregnant.
13. Patients or guardian able to sign informed consent.
14. No active CNS disease.
15. Platelet count > 100K.

Exclusion Criteria:

1) N/A

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2002-02-18 (Actual); Primary Completion 2006-05-19 (Actual); Study Completion 2006-05-19 (Actual)

PRIMARY OUTCOMES:
Response Rate | Within 180 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Donato, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T. M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson Cancer Center clinical trials web site — http://www.clinicaltrials.org